CLINICAL TRIAL: NCT00252005
Title: Protocol CV185017: A Phase 2 Randomized, Parallel-Arm Study of Oral Direct Factor Xa-Inhibitor Apixaban and Low Molecular Weight Heparin or Fondaparinux With A Vitamin K Antagonist In Subjects With Acute Symptomatic Deep-Vein Thrombosis
Brief Title: Oral Direct Factor Xa-inhibitor Apixaban in Patients With Acute Symptomatic Deep-vein Thrombosis-The Botticelli DVT Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV185-017
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2008-08

CONDITIONS: Deep-Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — apixaban

INTERVENTIONS:
Drug: Apixaban

SUMMARY:
The purpose of this clinical research study is to assess efficacy and safety of 3 doses of apixaban 5 mg twice a day, 10 mg twice a day and 20 mg once daily versus conventional treatment with low molecular weight heparin or fondaparinux and vitamin K antagonist in the treatment of subjects with acute symptomatic deep-vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing and able to give written informed consent.
2. Confirmed acute symptomatic DVT, i.e., proximal vein or extensive calf-vein thrombosis, involving at least the upper third part of the deep calf veins (trifurcation area) without concomitant symptomatic PE.
3. Women and men, ages 18 (or legal age of consent) to 90. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 1 week after the study in such a manner that the risk of pregnancy is minimized.

WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea for 12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35mIU/mL]. Even women who are using oral, implanted or, injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential. WOCBP must have negative serum or urine pregnancy test (minimum sensitivity 25IU/L or equivalent units of HCG) within 24 hours prior to the start of study medication.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Women with a positive pregnancy test on enrollment or prior to study drug administration.
3. More than 24 hours pre-randomization treatment with therapeutic dosages of unfractionated heparin (UFH), low molecular weight heparin (LMWH) or fondaparinux or more than a single starting dose of vitamin K antagonist (VKA) prior to randomization.
4. Uncontrolled hypertension: systolic blood pressure > 200 mm Hg or diastolic blood pressure > 110 mm Hg.
5. Creatinine clearance < 30 mL/min
6. Impaired liver function (ALT > 3 x ULN)
7. Use of ASA > 165 mg/day
8. WOCBP who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and for up to 1 week after the study.
9. Azole antifungals (e.g., ketoconazole), HIV protease inhibitors (e.g., ritonavir) and macrolide antibiotics (e.g., erythromycin).

NOTE: topical azole antifungal agents are permitted.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520
Dates: Start 2005-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The composite of symptomatic recurrent venous thromboembolism (i.e., recurrent deep-vein thrombosis or fatal or non-fatal pulmonary embolism and deterioration of the thrombotic burden as assessed by repeat bilateral
compression ultrasound and perfusion lung scan.

CONTACTS AND LOCATIONS:
Locations (72):
- United States (5):
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Chapel Hill, North Carolina
  - Local Institution, San Antonio, Texas
  - Local Institution, Fredericksburg, Virginia
  - Local Institution, Seattle, Washington
- Australia (9):
  - Local Institution, Garran, Australian Capital Territory
  - Local Institution, Caringbah, New South Wales
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Randwick, New South Wales
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, Clayton, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution, Perth, Western Australia
- Austria (2):
  - Local Institution, Graz
  - Local Institution, Vienna
- Czechia (7):
  - Local Institution, Hradec Králové
  - Local Institution, Karlovy Vary
  - Local Institution, Ostrava
  - Local Institution, Ostrava Poruba
  - Local Institution, Pilsen
  - Local Institution, Prague
  - Local Institution, Ústí nad Labem
- France (8):
  - Local Institution, Angers
  - Local Institution, Brest
  - Local Institution, Clermont-Ferrand
  - Local Institution, Créteil
  - Local Institution, Limoges
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Saint-Etienne
- Israel (9):
  - Local Institution, Afula
  - Local Institution, Ashkelon
  - Local Institution, Haifa
  - Local Institution, Holon
  - Local Institution, Jerusalem
  - Local Institution, Kfar Saba
  - Local Institution, Petah Tikva
  - Local Institution, Safed
  - Local Institution, Tel Aviv
- Italy (8):
  - Local Institution, Chieti
  - Local Institution, Milan
  - Local Institution, Padua
  - Local Institution, Pavia
  - Local Institution, Piacenza
  - Local Institution, Reggio Emilia
  - Local Institution, Treviso
  - Local Institution, Venezia
- Netherlands (6):
  - Local Institution, Amsterdam
  - Local Institution, Arnhem
  - Local Institution, Groningen
  - Local Institution, Hoofddorp
  - Local Institution, Maastricht
  - Local Institution, Zwolle
- Poland (7):
  - Local Institution, Bydgoszcz
  - Local Institution, Katowice
  - Local Institution, Krakow
  - Local Institution, Lublin
  - Local Institution, Poznan
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- South Africa (5):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Centurion, Gauteng
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Sunninghill, Gauteng
  - Local Institution, Somerset West, Western Cape
- Sweden (6):
  - Local Institution, Borås
  - Local Institution, Gothenburg
  - Local Institution, Halmstad
  - Local Institution, Jönköping
  - Local Institution, Stockholm
  - Local Institution, Västervik